CLINICAL TRIAL: NCT04550780
Title: Nation-wide Health Resource Consumption and Costs Associated With Mepolizumab (Nucala): a French SNDS Database Study
Brief Title: Nation-wide Health Resource Consumption and Costs Associated With Mepolizumab
Acronym: Resala
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0393
Record Dates: First submitted 2020-09-01; First posted 2020-09-16 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Asthma
Keywords: Mepolizumab
MeSH Terms: conditions — Asthma | interventions — mepolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The study population: The study population will comport all beneficiaries in the national French SNDS database who were prescribed mepolizumab and for whom health resource use data is available for the 12 months preceding and following a first filled prescription for mepolizumab.
  Interventions: Drug: Mepolizumab

INTERVENTIONS:
Drug: Mepolizumab — The first administration of mepolizumab.

SUMMARY:
Currently, no study has addressed real-life data describing changes in health resource consumption and related costs attributable to mepolizumab treatment. The aim of the current study is to fill this knowledge gap by performing an exhaustive extraction of data for patients receiving mepolizumab in the French single-payer health care system. The change in real-life health-resource usage and costs observed for these patients would provide the first evidence that mepolizumab is changing the care landscape for eligible severe asthma patients.

The overall objectives of this study are: (i) using the SNDS French national database, to identify a representative, nation-wide population of patients treated with mepolizumab with a follow-up period of at least 12 months, (ii) to describe the initial one-year changes in health resource use before and after the initiation of mepolizumab treatment and (iii) to estimate the change in associated costs for the first year of treatment. These initial data will additionally serve as a basis for the design of longer-term studies.

Primary objective: To estimate the change in associated costs for the first year of treatment

DETAILED DESCRIPTION:
Secondary objectives:

* To describe the initial one-year changes in health resource use before and after the initiation of mepolizumab treatment
* To further characterize rates of change in health resource usage and/or costs in subpopulations of interest (sex, age groups, severe asthma, uncontrolled asthma, COPD, diabetes)

This retrospective, non-interventional (not involving human subjects) database study will compare real-life patient health resource consumption before versus after a first injection of mepolizumab. Data concerning patients receiving mepolizumab will be collated for a 12-month period (the "baseline period") preceding a first index treatment (at "T0") and compared to a 12-month period occurring after the index treatment (the "exposure period").

ELIGIBILITY:
Inclusion Criteria:

* Beneficiary in the anonymous French national SNDS database
* The beneficiary received mepolizumab

Exclusion Criteria:

* Health resource use data covering the 12 months preceding the first filled prescription for mepolizumab are not available
* Health resource use data covering the time period starting at the first filled prescription for mepolizumab and ending at subsequent death or at 12 months later are not available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will comport all beneficiaries in the national French SNDS database who were prescribed mepolizumab and for whom health resource use data is available for the 12 months preceding and following a first filled prescription for mepolizumab.
Sampling Method: Probability Sample
Enrollment: 7938 (Actual)
Dates: Start 2021-12-03 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
The change in total health care costs for the year preceding the initiation of mepolizumab versus for the year after. | -12 months versus +12 months
  Cumulative per-beneficiary costs (including all health care resource uses and government benefits) will be described and contrasted between the baseline and exposure periods.
  Day 0 = the initiation of mepolizumab treatment.

SECONDARY OUTCOMES:
Change in drug consumption: mepolizumab | -12 months versus +12 months
  Drug consumption refers to the quantity of medication consumed.
Change in drug consumption: corticosteroids | -12 months versus +12 months
  Drug consumption refers to the quantity of medication consumed.
Change in drug consumption: asthma-specific medications | -12 months versus +12 months
  Drug consumption refers to the quantity of medication consumed.
Change in drug consumption: diabetes-related medications | -12 months versus +12 months
  Drug consumption refers to the quantity of medication consumed.
Change in the number of hospitalisations: all causes | -12 months versus +12 months
Change in the number of hospitalisations: asthma-related | -12 months versus +12 months
Change in the cumulative number of days of hospitalisation: all causes | -12 months versus +12 months
Change in the cumulative number of days of hospitalisation: asthma-related | -12 months versus +12 months
Change in the cumulative number of days of intensive care: all causes | -12 months versus +12 months
Change in the cumulative number of days of intensive care: asthma-related | -12 months versus +12 months
Change in the number of generalist consults | -12 months versus +12 months
  The cumulative numbers of consultations will be compared between the baseline and exposure period and differentiated according to type (general and specialist medical consults, nursing and other paramedical consults etc). Special attention will be given to pulmonology/allergology and metabolic/endocrine specialist consults, as well as nursing consults for injections.
Change in the number of specialist consults | -12 months versus +12 months
  The cumulative numbers of consultations will be compared between the baseline and exposure period and differentiated according to type (general and specialist medical consults, nursing and other paramedical consults etc). Special attention will be given to pulmonology/allergology and metabolic/endocrine specialist consults, as well as nursing consults for injections.
Change in the number of nursing consults | -12 months versus +12 months
  The cumulative numbers of consultations will be compared between the baseline and exposure period and differentiated according to type (general and specialist medical consults, nursing and other paramedical consults etc). Special attention will be given to pulmonology/allergology and metabolic/endocrine specialist consults, as well as nursing consults for injections.
Change in the number of other paramedical consults | -12 months versus +12 months
  The cumulative numbers of consultations will be compared between the baseline and exposure period and differentiated according to type (general and specialist medical consults, nursing and other paramedical consults etc). Special attention will be given to pulmonology/allergology and metabolic/endocrine specialist consults, as well as nursing consults for injections.
Change in the number of lung function assessments | -12 months versus +12 months
  Information concerning the laboratory and imaging assessments performed is available, but not their results. Special attention will be given to lung function, adrenal function, glycemia, and bone density assessments. The cumulative numbers of different assessments will be described and contrasted between the baseline and exposure periods.
Change in the number of adrenal function assessments | -12 months versus +12 months
  Information concerning the laboratory and imaging assessments performed is available, but not their results. Special attention will be given to lung function, adrenal function, glycemia, and bone density assessments. The cumulative numbers of different assessments will be described and contrasted between the baseline and exposure periods.
Change in the number of glycemia assessments | -12 months versus +12 months
  Information concerning the laboratory and imaging assessments performed is available, but not their results. Special attention will be given to lung function, adrenal function, glycemia, and bone density assessments. The cumulative numbers of different assessments will be described and contrasted between the baseline and exposure periods.
Change in the number of bone density assessments | -12 months versus +12 months
  Information concerning the laboratory and imaging assessments performed is available, but not their results. Special attention will be given to lung function, adrenal function, glycemia, and bone density assessments. The cumulative numbers of different assessments will be described and contrasted between the baseline and exposure periods.
The change in health care costs: mepolizumab | -12 months versus +12 months
  Cumulative per-beneficiary costs (including all health care resource uses and government benefits) will be described and contrasted between the baseline and exposure periods. This will be performed at several levels: (i) all costs regardless of source or potential link with diagnoses, (ii) costs due to mepolizumab, (iii) costs that can be associated with asthma-specific care, (iv) costs that can be associated with the monitoring and care for certain key comorbidities (diabetes, bone density/osteoporosis).
The change in health care costs: asthma-specific care | -12 months versus +12 months
  Cumulative per-beneficiary costs (including all health care resource uses and government benefits) will be described and contrasted between the baseline and exposure periods. This will be performed at several levels: (i) all costs regardless of source or potential link with diagnoses, (ii) costs due to mepolizumab, (iii) costs that can be associated with asthma-specific care, (iv) costs that can be associated with the monitoring and care for certain key comorbidities (diabetes, bone density/osteoporosis).
The change in health care costs: comorbidity care | -12 months versus +12 months
  Cumulative per-beneficiary costs (including all health care resource uses and government benefits) will be described and contrasted between the baseline and exposure periods. This will be performed at several levels: (i) all costs regardless of source or potential link with diagnoses, (ii) costs due to mepolizumab, (iii) costs that can be associated with asthma-specific care, (iv) costs that can be associated with the monitoring and care for certain key comorbidities (diabetes, bone density/osteoporosis).

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Molinari, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No
SNDS data are accessible only by specially trained and qualified individuals. Due to regulatory constraints, they cannot be made available to the public.

REFERENCES:
- See also: Resala on the Open Science Framework — https://osf.io/zg3us/